CLINICAL TRIAL: NCT00311012
Title: Dose-finding Study of SPP100 in Essential Hypertension
Brief Title: SPP100 Dose Finding Study in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A1201
Record Dates: First submitted 2006-03-31; First posted 2006-04-05 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: Hypertension, Aliskiren
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
This study will evaluate the efficacy of SPP100 in lowering blood pressure in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate essential hypertension
2. Age: ≥20 years old and <80 years old (at time informed consent obtained)
3. Sex: N/A
4. Admission status: Outpatient

Exclusion Criteria:

1. Pregnant women, lactating women, potentially pregnant women, or women who wish to become pregnant
2. Patients having a mean sitting diastolic blood pressure of ≥110 mmHg and/or a mean sitting systolic blood pressure of ≥180 mmHg at either Visit 2 or 3
3. Patients with secondary hypertension as a complication or patients suspected of having secondary hypertension(due to aortic coarctation, primary aldosteronism, coarctation of renal artery, renal hypertension
4. Patients suspected of having malignant hypertension

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2004-08; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure after 8 weeks
Diastolic blood pressure less than 90 mmHg or 10 mmHg or greater change from baseline after 8 weeks
Evaluate response to various doses by assessing the difference in mean sitting diastolic blood pressure after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Japan, Principal Investigator — Novartis Pharmaceuticals, Japan
Locations (1):
- Novartis Pharmaceuticals, Tokyo, Japan